CLINICAL TRIAL: NCT04164615
Title: A Randomized, Double-blind, Multi-center Phase Ⅲ Clinical Study to Evaluate the Recombinant Anti-HER2 Humanized Monoclonal Antibody or Placebo in Combination With Capecitabine for the Treatment of HER-2-positive Advanced Breast Cancer
Brief Title: Clinical Study of Recombinant Anti-HER2 Humanized Monoclonal Antibody (GB221) for Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENOR GB221-003；V1.1
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: HER-2-positive Advanced Breast Cancer
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB221+ Capecitabine tablets (Experimental): test drug+capecitabine
  Interventions: Drug: GB221
- Placebo control + capecitabine tablets (Placebo Comparator): placebo+capecitabine
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: GB221 — GB221:Lyophilized powder for injection; strength 110mg/bottle; the first administration of 8 mg/kg, intravenous drip for over 90 minutes; subsequently, the administration shall be given once every 3 weeks (one cycle), the dose is 6 mg/kg, intravenous drip for 30~90 minutes; The administration shall be continued until disease progression or presence of intolerable toxic reactions or subject's active withdrawal from clinical study.
  Capecitabine:Tablets; 500mg/tablet, 12 tablets/box; Total daily dose 2000 mg/m2, orally twice daily, one dose each in the morning and evening, administration for 2 weeks followed by a 1-week rest period, as a 3-week cycle. The administration shall be continued until disease progression or presence of intolerable toxic reactions or subject's active withdrawal from clinical study.
  Other Names: Capecitabine
  Arms: GB221+ Capecitabine tablets
Drug: Placebo control — Placebo control:Lyophilized powder for injection; strength 110mg/bottle; the first administration of 8 mg/kg, intravenous drip for over 90 minutes; subsequently, the administration shall be given once every 3 weeks (one cycle), the dose is 6 mg/kg, intravenous drip for 30~90 minutes; The administration shall be continued until disease progression or presence of intolerable toxic reactions or subject's active withdrawal from clinical study.
  Capecitabine:Tablets; 500mg/tablet, 12 tablets/box; Total daily dose 2000 mg/m2, orally twice daily, one dose each in the morning and evening, administration for 2 weeks followed by a 1-week rest period, as a 3-week cycle. The administration shall be continued until disease progression or presence of intolerable toxic reactions or subject's active withdrawal from clinical study.
  Other Names: capecitabine
  Arms: Placebo control + capecitabine tablets

SUMMARY:
The primary objective of this trial is to compare the progression-free survival (PFS) in two groups of combined therapy of GB221/ capecitabine tablets versus combined therapy of placebo/capecitabine tablets; the secondary objective is to evaluate the objective response rate (ORR),time to progression (TTP) from treatment period to week 12; overall survival (OS), safety, immunogenicity (anti-drug antibody), PFS of subjects during continued treatment period.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18 to 70 years;
2. Pathologically confirmed as advanced breast cancer and there is at least one measurable target lesion (based on RECIST V1.1):

   l According to Response Evaluation Criteria in Solid Tumors, the target lesions must be accurately measured in at least one dimension; l No previous radiotherapy, intervention for target lesions;
3. HER-2 positive [definition: including IHC (+++) or ISH positive; if IHC (++), HER-2 gene amplification detection should be further performed through fluorescence in situ hybridization (FISH) or chromogenic in situ hybridization (CISH),silver-enhanced in situ hybridization (SISH) and other methods. The test reports of the clinical study site associated with the subject should be provided];
4. The relapsed or metastatic patients who failed respond to the previous taxanes and/or anthracyclines, previous first-line chemotherapy for the metastatic lesion is acceptable;
5. The expected survival is 3 months or longer;
6. The function of major organs such as heart, liver and kidney are basically normal;
7. ECOG score ≤2;
8. Understand and voluntarily sign the written informed consent form;

2 Exclusion Criteria

1. Pregnant or breastfeeding females; or women of childbearing potential who have positive serum/urine pregnancy tests; females of childbearing potential and their partners are unwilling to adopt effective contraceptive methods during the clinical study period and within 6 months after the end of the study;
2. Received radiotherapy or chemotherapy within 4 weeks before randomization;
3. Received anti-tumor endocrine therapy within 2 weeks before randomization;
4. Previously received the standard anti-HER-2 treatment;
5. Previously received capecitabine treatment;
6. Subjects who previously received no taxanes; or subjects who respond to taxanes (no disease progression or intolerable toxic reactions);
7. The major organ function of subjects is abnormal. The laboratory test results are presented below:

Hematology test:

l Absolute neutrophil count (ANC) < 1.5×109/L; l Platelet count (PLT) <100×109/L; l Hemoglobin (Hb) < 90 g/L (no blood transfusion within 14 days);

Hepatic and renal function tests:

l Bilirubin (TBIL)>1.5×ULN (upper limit of normal); l Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)>2.5×ULN; if there is any hepatic metastasis, ALT and AST >5×ULN; l Serum creatinine (Cr) >1.5×ULN; 8. Left ventricular ejection fraction ( LVEF)<50%; 9. The organ system status of subjects:

1 Subjects with known or suspected brain metastasis: subjects with evidence indicating signs or symptoms of brain metastasis are not allowed to participate in this study unless such brain metastasis is excluded by CT or MRI. However, subjects whose brain metastasis lesions have been controlled can be enrolled (no progression within at least 4 weeks after radiotherapy and/or no neurological symptom or sign after surgical resection, treatment with dexamethasone or mannitol is not necessary);

1 Evidence showing severe or uncontrolled systemic diseases (e.g. unstable or non-compensated respiratory, cardiac, hepatic or renal disease);

1 Uncontrolled active infection (≥CTCAE grade 2); l Any other malignant tumor within 5 years, excluding patients with completely cured cervical in situ carcinoma or basal cell or squamous epithelial cell skin cancer);

1 Subjects who have any of the following cardiac conditions:

* Unstable angina pectoris;
* Medical history of congestive heart failure;
* Previous medical history of myocardial infarction, coronary artery bypass grafting or coronary stent implantation;
* Clinically significant pericardial diseases and valvular heart diseases;
* Cardiac arrhythmias requiring therapeutic intervention;
* Any other cardiac diseases which may cause safety risks for subjects if they are enrolled in this study; 1 Uncontrolled hypertension (defined as screening systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥110mmHg); 10. Immunodeficiency medical history, including positive HIV detection; 11. Positive hepatitis B surface antigen (HBsAg) and hepatitis B virus DNA of peripheral blood is not within the normal range; Positive hepatitis C virus antibody (HCV); 12. Subjects with drug abuse history or alcohol addiction history; 13. Participated in clinical study with drug intervention within one month before screening; 14. Subjects who are unsuitable for participation in this study at the discretion of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2016-11-24 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | through study completion, an average of 2 year
  To evaluate the efficacy of GB221 as defined by progression-free survival in patients with breast cancer.

SECONDARY OUTCOMES:
Objective Response Rate, ORR | through study completion, an average of 2 year
  To evaluate the efficacy of GB221 as defined by overall response rate, in patients with breast cancer.
Antidrug antibody, ADA | through study completion, an average of 2 year
  Antidrug antibody, ADA
Overall survival, OS | through study completion, an average of 2 year
  To evaluate the duration from the first administration to death because of any reason in patients with breast cancer.
PFS in the extended treatment phase | through study completion, an average of 2 year
  PFS in the extended treatment phase

CONTACTS AND LOCATIONS:
Locations (1):
- People's Liberation Army General Hospital The Fifth Medical Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No